CLINICAL TRIAL: NCT01483599
Title: A Phase 2 Multicenter, Randomized, Placebo- and Active-Comparator-Controlled, Dose-Ranging Trial to Evaluate CNTO 1959 for the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis (X-PLORE)
Brief Title: A Study to Evaluate CNTO 1959 in the Treatment of Patients With Moderate to Severe Plaque-type Psoriasis
Acronym: X-PLORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100673; CNTO1959PSO2001 (Other: Janssen Inc.); 2011-001066-17 (EudraCT Number)
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Psoriasis
Keywords: Moderate to Severe Plaque-Type Psoriasis; Psoriasis; Plaque-type psoriasis; CNTO 1959; adalimumab
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (7):
- CNTO 1959 (5 mg) (Experimental): CNTO 1959 5 mg at weeks 0, 4, and 16, then every 12 weeks through Week 40
  Interventions: Drug: CNTO 1959 (5 mg)
- CNTO 1959 (15 mg) (Experimental): CNTO 1959 15 mg at weeks 0, 8, and 16, then every 8 weeks through Week 40
  Interventions: Drug: CNTO 1959 (15 mg)
- CNTO 1959 (50 mg) (Experimental): CNTO 1959 50 mg at weeks 0, 4, and 16, then every 12 weeks through Week 40
  Interventions: Drug: CNTO 1959 (50 mg)
- CNTO 1959 (100 mg) (Experimental): CNTO 1959 100 mg at weeks 0, 8, and 16, then every 8 weeks through Week 40
  Interventions: Drug: CNTO 1959 (100 mg)
- CNTO 1959 (200 mg) (Experimental): CNTO 1959 200 mg at weeks 0, 4, and 16, then every 12 weeks through Week 40
  Interventions: Drug: CNTO 1959 (200 mg)
- Adalimumab (approved psoriasis dosing) (Active Comparator): Adalimumab 80 mg at week 0 followed by 40 mg at week 1 and every second week through Week 39 (i.e., Weeks 3, 5, 7, etc.)
  Interventions: Drug: Adalimumab
- Placebo to CNTO 1959 (100 mg) (Placebo Comparator): Placebo at weeks 0, 4, and 8; then crossover to CNTO 1959 100 mg at Week 16, then every 8 weeks through Week 40
  Interventions: Drug: CNTO 1959 (100 mg); Drug: Placebo

INTERVENTIONS:
Drug: CNTO 1959 (5 mg) — Subcutaneous (SC) injections
  Arms: CNTO 1959 (5 mg)
Drug: CNTO 1959 (15 mg) — SC injections
  Arms: CNTO 1959 (15 mg)
Drug: CNTO 1959 (50 mg) — SC injections
  Arms: CNTO 1959 (50 mg)
Drug: CNTO 1959 (100 mg) — SC injections
  Arms: CNTO 1959 (100 mg); Placebo to CNTO 1959 (100 mg)
Drug: CNTO 1959 (200 mg) — SC injections
  Arms: CNTO 1959 (200 mg)
Drug: Adalimumab — SC injections
  Arms: Adalimumab (approved psoriasis dosing)
Drug: Placebo — SC injections
  Arms: Placebo to CNTO 1959 (100 mg)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CNTO 1959 in the treatment of patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, dose-ranging study of CNTO 1959 in patients with moderate to severe plaque psoriasis. Patients who satisfy all inclusion and exclusion criteria will be assigned by chance to one of 7 treatment groups: a placebo group (a placebo is a treatment identical in appearance to CNTO 1959 but does not contain active drug), 1 of 5 dose groups for CNTO 1959, or adalimumab. Patients assigned to adalimumab will be dosed according to the labeled dosing for psoriasis. At Week 16, patients initially assigned to placebo will begin receiving CNTO 1959. Patients initially assigned to CNTO 1959 will continue to receive the same assigned dose level of study agent from Week 16 through Week 40. Patients receiving adalimumab will continue the labeled dosing regimen. All patients will be reassessed for clinical response every 4 weeks from Week 4 through Week 40. Patients will continue dosing through Week 40, with a subsequent efficacy and safety follow-up visit at Week 52. Patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque-type psoriasis with or without psoriatic arthritis for at least 6 months prior to first administration of any study agent
* Must be a candidate for phototherapy or systemic treatment for psoriasis (either new to treatment or having had previous treatment)
* Must be considered, in the opinion of the investigator, suitable candidates for adalimumab therapy
* If a woman, she must be postmenopausal, or if premenopausal, she must be either surgically sterile, practicing a highly effective method of birth control, or not heterosexually active during the study and for 5 months after receiving the last dose of study drug
* If a man, he must agree to use a double-barrier method of birth control (or must have been surgically sterilized) and to not donate sperm during the study and for 5 months after receiving the last dose of study drug.

Exclusion Criteria:

* History of or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Has a contra-indication to anti-TNF therapy
* Has a history of chronic or recurrent infectious disease
* Has a nonplaque form of psoriasis or has drug-induced psoriasis
* Has been previously treated with adalimumab
* Has received any therapeutic agent directly targeted to IL-12, IL-17, or IL-23, (including but not limited to ustekinumab, briakinumab [ABT-874], AIN457, and SCH900222) within 6 months of the first administration of study agent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2012-11-27 (Actual); Study Completion 2013-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (40):
- United States (18):
  - Birmingham, Alabama
  - Bakersfield, California
  - Los Angeles, California
  - Santa Monica, California
  - Ocala, Florida
  - Alpharetta, Georgia
  - Arlington Heights, Illinois
  - Skokie, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Andover, Massachusetts
  - Boston, Massachusetts
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Houston, Texas
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Canada (11):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Germany (4):
  - Hamburg
  - Mahlow
  - Münster
  - Schwerin
- Poland (4):
  - Gdansk
  - Gmina Końskie
  - Lodz
  - Wroclaw

REFERENCES:
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Gordon KB, Duffin KC, Bissonnette R, Prinz JC, Wasfi Y, Li S, Shen YK, Szapary P, Randazzo B, Reich K. A Phase 2 Trial of Guselkumab versus Adalimumab for Plaque Psoriasis. N Engl J Med. 2015 Jul 9;373(2):136-44. doi: 10.1056/NEJMoa1501646. PMID 26154787

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (CP): Participants received placebo matched to CNTO1959 subcutaneous injection at Week 0, Week 4 and Week 8.
- CNTO1959 5 mg (CP): Participants received CNTO1959 5 milligram (mg) subcutaneous injection at Week 0 and Week 4 and matching placebo subcutaneous injection at Week 8.
- CNTO1959 15 mg (CP): Participants received CNTO1959 15 mg subcutaneous injection at Week 0 and Week 8 and matching placebo subcutaneous injection at Week 4.
- CNTO1959 50 mg (CP): Participants received CNTO1959 50 mg subcutaneous injection at Week 0 and Week 4 and matching placebo subcutaneous injection at Week 8.
- CNTO1959 100 mg (CP): Participants received CNTO1959 100 mg subcutaneous injection at Week 0 and Week 8 and matching placebo subcutaneous injection at Week 4.
- CNTO1959 200 mg (CP): Participants received CNTO1959 200 mg subcutaneous injection at Week 0 and Week 4 and matching placebo subcutaneous injection at Week 8.
- Adalimumab (CP): Participants received Adalimumab 80 mg subcutaneous injection at Week 0 and 40 mg at Week 1 and every other week up to Week 15.
- Placebo -> 100 mg CNTO1959 (After CP): Same participants who received placebo and completed controlled period transitioned to receive 100 mg CNTO1959 at Week 16 and once in every 8 weeks through Week 40.
- CNTO1959 5 mg (After CP): Participants who received CNTO1959 5 mg and completed controlled period continued to receive CNTO1959 5 mg starting at Week 16 and once in every 12 weeks through Week 40.
- CNTO1959 15 mg (After CP): Participants who received CNTO1959 15 mg and completed controlled period continued to receive CNTO1959 15 mg starting at Week 16 and once in every 8 weeks through Week 40.
- CNTO1959 50 mg (After CP): Participants who received CNTO1959 50 mg and completed controlled period continued to receive CNTO1959 50 mg starting at Week 16 and once in every 12 weeks through Week 40.
- CNTO1959 100 mg (After CP): Participants who received CNTO1959 100 mg and completed controlled period continued to receive CNTO1959 100 mg starting at Week 16 and once in every 8 weeks through Week 40.
- CNTO1959 200 mg (After CP): Participants who received CNTO1959 200 mg and completed controlled period continued to receive CNTO1959 200 mg starting at Week 16 and once in every 12 weeks through Week 40.
- Adalimumab (After CP): Participants who received adalimumab and completed controlled period continued to receive adalimumab 40 mg starting at week 17 and every other week thereafter through Week 39.
Period: Controlled Period (CP) (up to Week 16)
Arm/Group | Placebo (CP) | CNTO1959 5 mg (CP) | CNTO1959 15 mg (CP) | CNTO1959 50 mg (CP) | CNTO1959 100 mg (CP) | CNTO1959 200 mg (CP) | Adalimumab (CP) | Placebo -> 100 mg CNTO1959 (After CP) | CNTO1959 5 mg (After CP) | CNTO1959 15 mg (After CP) | CNTO1959 50 mg (After CP) | CNTO1959 100 mg (After CP) | CNTO1959 200 mg (After CP) | Adalimumab (After CP)
Started | 42 | 41 | 41 | 42 | 42 | 42 | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 42 | 41 | 41 | 42 | 42 | 41 | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 39 | 38 | 41 | 39 | 40 | 38 | 39 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 0 | 3 | 2 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 1 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: After Controlled Period(Week 16-Week 40)
Arm/Group | Placebo (CP) | CNTO1959 5 mg (CP) | CNTO1959 15 mg (CP) | CNTO1959 50 mg (CP) | CNTO1959 100 mg (CP) | CNTO1959 200 mg (CP) | Adalimumab (CP) | Placebo -> 100 mg CNTO1959 (After CP) | CNTO1959 5 mg (After CP) | CNTO1959 15 mg (After CP) | CNTO1959 50 mg (After CP) | CNTO1959 100 mg (After CP) | CNTO1959 200 mg (After CP) | Adalimumab (After CP)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 38 | 41 | 39 | 40 | 38 | 39
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 29 | 37 | 37 | 39 | 35 | 32
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 4 | 2 | 1 | 3 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population analyzed included all participants who were randomized.
Groups:
- Placebo: Participants received placebo matched to CNTO1959 subcutaneous injection at Week 0, Week 4, Week 8 then 100 mg CNTO1959 at Week 16 and once every 8 weeks thereafter through Week 40.
- CNTO1959 5 mg: Participants received CNTO1959 5 milligram (mg) subcutaneous injection at Week 0, Week 4 and once every 12 weeks thereafter through Week 40.
- CNTO1959 15 mg: Participants received CNTO1959 15 mg subcutaneous injection at Week 0, Week 8 and once every 8 weeks thereafter through Week 40.
- CNTO1959 50 mg: Participants received CNTO1959 50 mg subcutaneous injection at Week 0, Week 4 and once every 12 weeks thereafter through Week 40.
- CNTO1959 100 mg: Participants received CNTO1959 100 mg subcutaneous injection at Week 0, Week 8 and once every 8 weeks thereafter through Week 40.
- CNTO1959 200 mg: Participants received CNTO1959 200 mg subcutaneous injection at Week 0, Week 4 and once every 12 weeks thereafter through Week 40.
- Adalimumab: Participants received Adalimumab 80 mg subcutaneous injection at Week 0, 40 mg at Week 1 and once every other week thereafter through Week 39.
- Total: Total of all reporting groups
Arm/Group | Placebo | CNTO1959 5 mg | CNTO1959 15 mg | CNTO1959 50 mg | CNTO1959 100 mg | CNTO1959 200 mg | Adalimumab | Total
Number analyzed (Participants) | 42 | 41 | 41 | 42 | 42 | 42 | 43 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 41 | 39 | 39 | 41 | 36 | 40 | 35 | 271
  >=65 years | 1 | 1 | 2 | 1 | 6 | 2 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.97) | 45.2 (13.92) | 43.8 (13.5) | 42.6 (12.14) | 45.3 (13.72) | 45.1 (10.96) | 47.5 (14.91) | 44.9 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 13 | 12 | 10 | 11 | 13 | 86
  Male | 28 | 28 | 28 | 30 | 32 | 31 | 30 | 207
Region of Enrollment [Number; unit: participants]
  Germany | 2 | 2 | 4 | 5 | 4 | 3 | 3 | 23
  Belgium | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 5
  Poland | 7 | 8 | 7 | 10 | 7 | 8 | 8 | 55
  Canada | 13 | 11 | 11 | 11 | 12 | 14 | 11 | 83
  United States | 18 | 19 | 19 | 16 | 18 | 16 | 21 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 16
Description: PGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point. Lesions were graded as erythema [0 (no evidence of plaque) to 5 (dusky to deep red coloration)], induration [0 (no plaque evaluation) to 5 (marked plaque evaluation)] and scaling [0 (no evidence of scaling) to 5 (severe; very thick tenacious scaling)]. The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0= cleared; 1= minimal; 2= mild; 3= moderate; 4= marked and 5= severe).
Time Frame: Week 16
Population: Population analyzed included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CNTO1959 5 mg | CNTO1959 15 mg | CNTO1959 50 mg | CNTO1959 100 mg | CNTO1959 200 mg | Adalimumab
Number analyzed (Participants) | 42 | 41 | 41 | 42 | 42 | 42 | 43
percentage of participants | 7.1 | 34.1 | 61.0 | 78.6 | 85.7 | 83.3 | 58.1
Statistical Analysis 1: Comparison: Placebo vs CNTO1959 5 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (less than or equal to (<=) 90 kilogram (kg), greater than (>) 90 kg); Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 2: Comparison: Placebo vs CNTO1959 15 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 50 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 100 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 5: Comparison: Placebo vs CNTO1959 200 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 6: Comparison: Placebo vs Adalimumab; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

2. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. PASI 75 response was defined as at least a 75% reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: Population analyzed included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CNTO1959 5 mg | CNTO1959 15 mg | CNTO1959 50 mg | CNTO1959 100 mg | CNTO1959 200 mg | Adalimumab
Number analyzed (Participants) | 42 | 41 | 41 | 42 | 42 | 42 | 43
percentage of participants | 4.8 | 43.9 | 75.6 | 81.0 | 78.6 | 81.0 | 69.8
Statistical Analysis 1: Comparison: Placebo vs CNTO1959 5 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 2: Comparison: Placebo vs CNTO1959 15 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 50 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 100 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 5: Comparison: Placebo vs CNTO1959 200 mg; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test
Statistical Analysis 6: Comparison: Placebo vs Adalimumab; p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by baseline weight (<=90 kg, >90 kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

3. Secondary Outcome: Difference in Percentage of Participants With Physician Global Assessment (PGA) Score of Cleared (0) or Minimal (1) in CNTO1959 Groups Compared With Adalimumab Group at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: Population analyzed included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | CNTO1959 5 mg | CNTO1959 15 mg | CNTO1959 50 mg | CNTO1959 100 mg | CNTO1959 200 mg | Adalimumab
Number analyzed (Participants) | 41 | 41 | 42 | 42 | 42 | 43
percentage of participants | 34.1 | 61.0 | 78.6 | 85.7 | 83.3 | 58.1
Statistical Analysis 1: Comparison: CNTO1959 5 mg vs Adalimumab; The difference in percentage was calculated as the percentage of CNTO 1959 participants achieving a PGA score of cleared (0) or minimal (1) minus percentage of adalimumab participants achieving a PGA score of cleared (0) or minimal (1); Test type: Superiority or Other; Difference in Percentage = -24.0, 95% CI 2-sided [-44.0 to -4.0]
Statistical Analysis 2: Comparison: CNTO1959 15 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 2.8, 95% CI 2-sided [-17.9 to 23.5]
Statistical Analysis 3: Comparison: CNTO1959 50 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 20.4, 95% CI 2-sided [1.5 to 39.3]
Statistical Analysis 4: Comparison: CNTO1959 100 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 27.7, 95% CI 2-sided [9.8 to 45.6]
Statistical Analysis 5: Comparison: CNTO1959 200 mg vs Adalimumab; Test type: Superiority or Other; Difference in Percentage = 25.4, 95% CI 2-sided [7.2 to 43.6]

4. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 40
Description: as for outcome 1
Time Frame: Week 40
Population: Population analyzed included all participants who were randomized. Here, 'Number of participants analyzed' signifies those participants who were evaluable for this outcome measure. The placebo reporting group was not planned to be analyzed in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | CNTO1959 5 mg | CNTO1959 15 mg | CNTO1959 50 mg | CNTO1959 100 mg | CNTO1959 200 mg | Adalimumab
Number analyzed (Participants) | 34 | 37 | 38 | 39 | 37 | 37
percentage of participants | 35.3 | 59.5 | 71.1 | 76.9 | 81.1 | 48.6
Statistical Analysis 1: Comparison: CNTO1959 5 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = -15.4, 95% CI 2-sided [-37.7 to 6.9]
Statistical Analysis 2: Comparison: CNTO1959 15 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 10.8, 95% CI 2-sided [-10.7 to 32.4]
Statistical Analysis 3: Comparison: CNTO1959 50 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 22.7, 95% CI 2-sided [1.8 to 43.6]
Statistical Analysis 4: Comparison: CNTO1959 100 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 28.7, 95% CI 2-sided [8.5 to 49.0]
Statistical Analysis 5: Comparison: CNTO1959 200 mg vs Adalimumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Difference in Percentage = 32.9, 95% CI 2-sided [13.0 to 52.8]

5. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants.
Time Frame: Baseline and Week 16
Population: Population analyzed included all participants who were randomized. Here, 'Number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CNTO1959 5 mg | CNTO1959 15 mg | CNTO1959 50 mg | CNTO1959 100 mg | CNTO1959 200 mg | Adalimumab
Number analyzed (Participants) | 42 | 39 | 41 | 40 | 40 | 39 | 39
units on a scale | -2.3 (6.80) | -6.2 (5.24) | -10.3 (5.49) | -11.1 (7.38) | -10.8 (7.34) | -11.4 (6.83) | -10.1 (9.00)
Statistical Analysis 1: Comparison: Placebo vs CNTO1959 5 mg; Test type: Superiority or Other; p = 0.008, ANOVA on the van Der Waerden score
Statistical Analysis 2: Comparison: Placebo vs CNTO1959 15 mg; Test type: Superiority or Other; p < 0.001, ANOVA on the van Der Waerden score
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 50 mg; Test type: Superiority or Other; p < 0.001, ANOVA on the van Der Waerden score
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 100 mg; Test type: Superiority or Other; p < 0.001, ANOVA on the van Der Waerden score
Statistical Analysis 5: Comparison: Placebo vs CNTO1959 200 mg; Test type: Superiority or Other; p < 0.001, ANOVA on the van Der Waerden score
Statistical Analysis 6: Comparison: Placebo vs Adalimumab; Test type: Superiority or Other; p < 0.001, ANOVA on the van Der Waerden score

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) up to Week 52
Description: Safety analysis set included all randomized participants who received at least 1 injection of study treatment (partial or complete).
Arm/Group | Placebo (CP) | CNTO1959 5 mg (CP) | CNTO1959 15 mg (CP) | CNTO1959 50 mg (CP) | CNTO1959 100 mg (CP) | CNTO1959 200 mg (CP) | Adalimumab (CP) | Placebo -> 100 mg CNTO1959 (After CP) | CNTO1959 5 mg (After CP) | CNTO1959 15 mg (After CP) | CNTO1959 50 mg (After CP) | CNTO1959 100 mg (After CP) | CNTO1959 200 mg (After CP) | Adalimumab (After CP)
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/41 | 0/41 | 3/42 | 0/42 | 0/41 | 1/43 | 0/39 | 2/38 | 0/41 | 0/39 | 2/40 | 0/38 | 1/38
Other Adverse Events (participants affected / at risk) | 13/42 | 15/41 | 10/41 | 10/42 | 7/42 | 8/41 | 10/43 | 16/39 | 12/38 | 4/41 | 11/39 | 16/40 | 12/38 | 13/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=42) | CNTO1959 5 mg (CP) (N=41) | CNTO1959 15 mg (CP) (N=41) | CNTO1959 50 mg (CP) (N=42) | CNTO1959 100 mg (CP) (N=42) | CNTO1959 200 mg (CP) (N=41) | Adalimumab (CP) (N=43) | Placebo -> 100 mg CNTO1959 (After CP) (N=39) | CNTO1959 5 mg (After CP) (N=38) | CNTO1959 15 mg (After CP) (N=41) | CNTO1959 50 mg (After CP) (N=39) | CNTO1959 100 mg (After CP) (N=40) | CNTO1959 200 mg (After CP) (N=38) | Adalimumab (After CP) (N=38)
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=42) | CNTO1959 5 mg (CP) (N=41) | CNTO1959 15 mg (CP) (N=41) | CNTO1959 50 mg (CP) (N=42) | CNTO1959 100 mg (CP) (N=42) | CNTO1959 200 mg (CP) (N=41) | Adalimumab (CP) (N=43) | Placebo -> 100 mg CNTO1959 (After CP) (N=39) | CNTO1959 5 mg (After CP) (N=38) | CNTO1959 15 mg (After CP) (N=41) | CNTO1959 50 mg (After CP) (N=39) | CNTO1959 100 mg (After CP) (N=40) | CNTO1959 200 mg (After CP) (N=38) | Adalimumab (After CP) (N=38)
Fatigue (General disorders) | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injection Site Erythema (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 6 | 4 | 1 | 1 | 2 | 2 | 4 | 6 | 1 | 7 | 4 | 5 | 6
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 3 | 2 | 4 | 4 | 1 | 0 | 3 | 2 | 3
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 3 | 2 | 0 | 0 | 1 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 4 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.